CLINICAL TRIAL: NCT06288243
Title: Examination Of The Correlation Between Functionality And Cognition And Swallowing Skills In Patients With Acute Stroke
Brief Title: Functionality, Cognition And Swallowing Skills In Patients With AcuteSTROKE
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hilal Berber Çiftci, PhD Lecturer, Medipol University
Other Study IDs: Samatya
Record Dates: First submitted 2024-02-15; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Stroke, Acute; Swallowing Disorder; Cognitive Impairment; Stroke; Movement Disorders; Dysphagia
Keywords: stroke; acute stroke; dysphagia; cognitive status; functionality
MeSH Terms: conditions — Stroke; Deglutition Disorders; Cognitive Dysfunction; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Clinician-observed assessment tests — Turkish Modified Mann Swallowing Ability Test, which evaluates swallowing skills Standardized Mini-Mental Test assessing Cognitive Status Modified Rankin Scale to evaluate functionality

SUMMARY:
Aim: Studies in which the results of the screening test evaluating swallowing skills in acute stroke patients are evaluated together with other components that may affect swallowing function are limited. The aim of this study is to determine which factors are associated with swallowing abilities in patients with acute stroke, including lesion location, cognitive level, clinical features, risk factors for stroke, and level of functionality.

Methods: The 97 acute stroke patients included in the study were grouped in terms of lesion type, affected side, and risk factors for stroke. Turkish MMASA (TR-MMASA) was used to evaluate the swallowing ability of the patients. Additionally, Standardized Mini Mental Test (SMMT) and Modified Rankin Scale (MRS) were applied to evaluate cognition level and functionality, respectively.

DETAILED DESCRIPTION:
Dysphagia after acute stroke is common in the early stage and risk factors should be defined by actively evaluating it. Studies in which the results of the screening test evaluating swallowing skills in acute stroke patients are evaluated together with other components that may affect swallowing function are limited. The aim of this study is to determine which factors are associated with swallowing abilities in patients with acute stroke, including lesion location, cognitive level, clinical features, risk factors for stroke, and level of functionality. We evaluated the pre-swallowing skills of stroke patients with the Turkish translation of MMASA, a current screening test (TR-MMASA). We focused on the fact that the level of functionality and cognition may also be low in acute stroke patients with a high risk of swallowing disorders. We also investigated the consistency of the TR-MMASA swallowing screening test, which we assumed might be compatible with other tests evaluating cognition and functionality.

The 97 acute stroke patients included in the study were grouped in terms of lesion type, affected side, and risk factors for stroke. Inclusion criteria were a stroke diagnosis by a specialist neurologist with radiological confirmation cranial computed tomography (CT) or magnetic resonance imaging. Exclusion criteria were a history of head and neck cancer or trauma, having received radiotherapy in the last 12 months, a neurological or neurodegenerative disorder independent of stroke affecting swallowing function. Data collection was completed by completing the Turkish MMASA(TR-MMASA) dysphagia screening test, Standardized Mini Mental Test (SMMT) and Modified Rankin Scale (MRS) and demographic information forms. In the demographic information form, information about the participants' age, gender, lesion type, affected side, time spent after stroke, dominant side, and education level were recorded.

The study protocol was approved by the Istanbul Medipol University Non-Invasive Clinical Research Ethics Committee (Decree No: 124).Written permission was obtained from Istanbul Training and Research Hospital Neurology Clinic to conduct the study. Written and verbal consent was obtained from the patients through an informed consent form to participate in the study. The consent of the patients who were unable to give consent was obtained from their first-degree relatives. The study was conducted in accordance with the Principles of the Declaration of Helsinki.

SPSS (Statistical Package for the Social Sciences Inc; Chicago, IL, USA) 24.0 statistical package program was used to analyze the data. Descriptive statistics (number-percentage ratios, mean values, standard deviation value, median, minimum-maximum values) were used to express the data obtained in the study. Chi-square test technique was applied to determine whether there is dependency between the variables. ANOVA test was used to determine whether there is a dependency between more than two variables. Confidence interval was accepted as 95% (p<0.05) in statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Stroke diagnosis by a specialist neurologist with radiological confirmation cranial computed tomography (CT) or magnetic resonance imaging

Exclusion Criteria:

* History of head and neck cancer or trauma,
* Having received radiotherapy in the last 12 months,
* A neurological or neurodegenerative disorder independent of stroke affecting swallowing function.

Ages: 45 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had an acute stroke and were treated in the neurology clinic
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
The Correlation Between Swallowing Skills and Cognitive Status | During the first 5 months of the study.
  Is there correlation between the scores obtained from the TR-MMASA(Turkish Modified Mann Swallowing Ability test and the scores obtained from the SMMT(Standardized Mini Mental Test)? The TR-MMASA test is a test based on clinical observation that gives a score between 92 and 100 for the patient's swallowing skills. A score of 92 and below means non-oral nutrition, and a score above 92 means that it can be fed orally.
  SMMT test is a test that measures the cognitive level of the patient based on clinical observation between 0-30. As the score value decreases, it means that the cognitive level worsens.
The Correlation Between Swallowing Skills and Functionality | During the first 5 months of the study.
  Is there correlation between the scores obtained from the TR-MMASA(Turkish Modified Mann Swallowing Ability) test and the scores obtained from the MRS(Modified Rankin Scale) test? The TR-MMASA test is a test based on clinical observation that gives a score between 92 and 100 for the patient's swallowing skills. A score of 92 and below means non-oral nutrition, and a score above 92 means that it can be fed orally.
  MRS test is the test that evaluates the patient's functional independence. Scoring 0-2 points from the test means that the patient is functionally dependent, and scoring 3-6 points means that the patient is functionally independent.

SECONDARY OUTCOMES:
The relationship between stroke risk factors and swallowing skills | During the first 5 months of the study.
  Is there a significant relationship between TR-MMASA(Turkish Modified Mann Swallowing Ability) test scores and stroke risk factors (low, medium, high)?
The relationship between demographic informations and swallowing skills | During the first 5 months of the study.
  Is there a significant relationship between the scores obtained from the TR-MMASA test and demographic information (age, gender, lesion type(ischemic-hemorragic), affected side(right-left-no motor deficit))?

CONTACTS AND LOCATIONS:
Overall Officials: Seyhun Topbaş, Prof.Dr., Study Director — Medipol University
Locations (1):
- Medipol University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carnaby-Mann G, Lenius K. The bedside examination in dysphagia. Phys Med Rehabil Clin N Am. 2008 Nov;19(4):747-68, viii. doi: 10.1016/j.pmr.2008.05.008. PMID 18940639
- [Result] Antonios N, Carnaby-Mann G, Crary M, Miller L, Hubbard H, Hood K, Sambandam R, Xavier A, Silliman S. Analysis of a physician tool for evaluating dysphagia on an inpatient stroke unit: the modified Mann Assessment of Swallowing Ability. J Stroke Cerebrovasc Dis. 2010 Jan;19(1):49-57. doi: 10.1016/j.jstrokecerebrovasdis.2009.03.007. PMID 20123227